CLINICAL TRIAL: NCT07306481
Title: The Efficacy of Preoperative Oral Administration of Lactobacillus Reuteri Combined With Preoperative Neoadjuvant/Conversion Immunotherapy in Patients With Primary Resectable Liver Cancer: a Prospective Study
Brief Title: The Efficacy of Preoperative Oral Administration of Lactobacillus Reuteri Combined With Preoperative Neoadjuvant/Conversion Immunotherapy in Patients With Primary Resectable Liver Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LRHCC-2025
Record Dates: First submitted 2025-11-22; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: HCC - Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lr group (Experimental)
  Interventions: Dietary Supplement: Dietary Supplement: L. reuteri DSM 17938
- Con group (No Intervention)

INTERVENTIONS:
Dietary Supplement: Dietary Supplement: L. reuteri DSM 17938 — 1 * 10^8 CFU of L. reuteri DSM 17938 two capsules per day for 3 months
  Arms: Lr group

SUMMARY:
On the basis of previous studies, this study intends to explore the efficacy of preoperative oral administration of Lactobacillus reuteri (Lr) combined with preoperative neoadjuvant/conversion therapy in patients with primary resectable hepatocellular carcinoma (HCC). We hypothesize that this combination represents a novel, microbiota-based therapeutic strategy to facilitate perioperative hepatic recovery and improve long-term survival outcomes.

This study is an open-label, randomized, blank-controlled clinical trial. Patients undergoing liver resection were randomly allocated to one of two groups. The intervention group received preoperative oral Lactobacillus reuteri (Lr) supplementation alongside neoadjuvant/conversion immunotherapy. The control group received preoperative neoadjuvant/conversion immunotherapy alone. Fecal and peripheral blood samples will be collected at baseline (pre-medication), 3 days prior to surgery, and at 5 days, 1, 3, 6, 9, 12, 18, and 24 months postoperatively. Intraoperative liver tissue samples will also be obtained. Statistical analyses will be performed to compare intergroup differences in postoperative liver function recovery, overall survival, hepatic and peripheral immune markers, and gut microbiota composition.

This study aims to develop adjuvant strategies to enhance therapeutic outcomes for HCC patients undergoing preoperative neoadjuvant/conversion immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Understanding and voluntarily signing the informed consent form for this study;
2. Age≥18 years and ≤75 years; gender not restricted;
3. Histologically (pathologically), cytologically, or radiologically confirmed hepatocellular carcinoma (HCC);
4. Patients who require preoperative immune checkpoint inhibitor (ICI) combination therapy followed by potentially curative hepatectomy;
5. No prior systemic therapy for HCC, including chemotherapy, targeted therapy, or immunotherapy had been administered before enrollment.;
6. Patients with a history of prior curative surgery or curative ablation are allowed, except for those with recurrence within 2 years post-curative treatment or prior receipt of other local therapies;
7. At least one measurable lesion meets RECIST v1.1 criteria;
8. Child-Pugh liver function rating: grade A or B;
9. The expected survival period is greater than 3 months;
10. Patients must be able to take food orally independently;
11. Preoperative ECOG physical condition score 0-1 points;
12. Normal coagulation function, no activebleeding or thrombotic diseases; A. International standardized ratio INR≤1.5×ULN; B. Partial thromboplastin time APTT≤1.5×ULN;
13. Has adequate organ and bone marrow function, laboratory test values within 7 days prior to enrollment meet the following requirements (no blood components, cell growth factors, albumin, or other corrective drugs are allowed within 14 days prior to laboratory test), as follows: 1) Blood routine: absolute neutrophil count≥1.5×109/L; platelet count≥75×109/L; hemoglobin conten≥9.0 g/dL. 2) Liver function: serum total bilirubin≤2× upper limit of normal value (ULN); alanine aminotransferase and aspartate transferas≤5×ULN; Serum albumin ≥28 g/L; alkaline phosphatase≤5×ULN. 3) Renal function: serum creatinine≤1.5×ULN or clearance of creatinine≥50mL/min(Cockcroft-Gault formula); Urine routine results showed that urine protein <2+; For patients with urine protein ≥2+ on routine urine tests at baseline, 24-hour urine collection and 24-hour protein quantification <1g should be performed.

Exclusion Criteria:

1. Inability to comply with the study protocols or procedures;
2. Known intrahepatic cholangiocarcinoma, sarcomatoid hepatocellular carcinoma, mixed cell carcinoma (ICC more than 30%) and fibrolaminar cell carcinoma
3. Hepatic encephalopathy, hepatorenal syndrome, or severe decompensated cirrhosis;
4. Planned use of probiotics, yogurt, or bacterial-fortified foods during the treatment period;
5. Use of probiotics or antibiotic within 2 months before the trial;
6. Patients with severe mental illness;
7. Patients under fasting or fluid restriction (e.g., complete bowel obstruction, active gastrointestinal bleeding, etc.);
8. Patients with chronic digestive system diseases, such as irritable bowel syndrome, malabsorption syndrome, inflammatory bowel disease, or ileostomy;
9. Allergy to the trial product or its components, inability to swallow tablets, unwillingness or inability to receive intravenous administration, or a history of severe infusion-related reactions to monoclonal antibodies or any other active malignancies during the initial study treatment administration;
10. Participants in other drug, dietary supplement, probiotic, or prebiotic clinical studies within the past 1 months prior to enrollment
11. Pregnant or lactating women;
12. History of other malignancies within the past 5 years, except for completely resected basal cell carcinoma or squamous cell carcinoma of the skin, or cervical carcinoma in situ;
13. Any medical or non-medical condition that the researcher deems unsuitable for participation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12-20 (Estimated); Primary Completion 2028-06-20 (Estimated); Study Completion 2028-12-20 (Estimated)

PRIMARY OUTCOMES:
Comparison of liver function recovery with ALT and AST | 5 days, 1 month, 3 months, 6 months, 9 months, 12 months, 18 months, and 24 months after surgery
  The levels of the alanine aminotransferase (ALT) and aspartate aminotransferase (ALT) after surgery will be compared.
Comparison of liver function recovery with total bilirubin | 5 days, 1 month, 3 months, 6 months, 9 months, 12 months, 18 months, and 24 months after surgery
  The levels of the total bilirubin after surgery will be compared.
Comparison of liver function recovery with prothrombin activity | 5 days, 1 month, 3 months, 6 months, 9 months, 12 months, 18 months, and 24 months after surgery
  The levels of the prothrombin after surgery will be compared.
Incidence of postoperative complications | 30 days after the surgery
  The postoperative complication rates including surgical site infection, hemorrhage, and bile leakage.

SECONDARY OUTCOMES:
Analysis of hepatic tissue microbiota | During surgery
  Postoperative liver specimens will be collected to compare or quantitatively detect microbial content (e.g., Lactobacillus reuteri) in liver tissues (tumor and peritumoral regions) through culture-based methods, or to assess microbial community diversity changes via microbiome sequencing.
Alterations in gut microbiota | Before intervention, 3 days before surgery, and 5 days, 1 month, 3 months, 6 months, 9 months, 12 months, 18 months, and 24 months after surgery
  16S rRNA sequencing will be used to measure fecal sample. The alpha and beta diversity of gut microbiota between two groups will be analyzed, including a series of statistical analysis indexes such as Chao, Shannon, Simpsonace, Simpson and Coverage, in order to reflect the microbial community diversity.
Differences among hepatic immune cell subsets | During surgery
  Single-cell sequencing will be used to analyzed the immune cell subsets in tumor tissues and paired normal tissues. The immune cell clusters comprised: 9 clusters of CD4+ T cells (CD3+CD4+), 8 clusters of CD8+ T cells (CD3+CD8+), 3 clusters of B cells (CD3-CD19+), 2 clusters of monocytes (CD3-CD19-CD14+) and 10 clusters of other subsets, such as dendritic cells (DCs, CD3-CD19-CD14-CD20-HLA-DR+), and NK cells (CD3-CD19-CD14-C-D20-CD56+).
The alterations of peripheral immune cell subsets | 3 days before surgery, and 1, 3, 6, 9, 12, 18, and 24 months after surgery
  Single-cell sequencing will be used to analyze the immune cell subsets in peripheral blood. The peripheral immune cell subsets comprised: 9 clusters of CD4+ T cells (CD3+CD4+), 8 clusters of CD8+ T cells (CD3+CD8+), 3 clusters of B cells (CD3-CD19+), 2 clusters of monocytes (CD3-CD19-CD14+) and 10 clusters of other subsets, such as dendritic cells (DCs, CD3-CD19-CD14-CD20-HLA-DR+), and NK cells (CD3-CD19-CD14-C-D20-CD56+).
The alterations of immune cytokines | 3 days before surgery, and 1, 3, 6, 9, 12, 18, and 24 months after surgery
  Standardized luminex-based multiplex bead technology or elisa assay will be used to assess the dynamic changes of immune cytokines at key time points. The immune cytokines included TNF-α, IFN-γ, CXCL10, G-CSF, IL-1β, IL-1RA, IL-2, IL-4, IL-5, IL-6, IL-7, IL-8, IL-9, IL-10, IL-12p70, IL-13, IL-15, IL-17, PDGF-BB, MCP-1, MIP-1α, MIP-1β, GM-CSF, eotaxin, FGF, and RANTES.
Potential impact on long-term postoperative survival | 1year and 2year
  1-year and 2-year recurrence-free survival (RFS) and overall survival (OS) rate。